CLINICAL TRIAL: NCT05959044
Title: Effect of Folic Acid on Motor Aspects of Daily Living and Oxidative Stress in Levodopa Treated Parkinson's Disease Patients: A Randomized, Double-Blind, Placebo Controlled Trial
Brief Title: Effect of Folic Acid in Levodopa Treated Parkinson's Disease Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Shimu Akter Ayshi, MD Resident, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BSMMU/2023/6247
Record Dates: First submitted 2023-07-15; First posted 2023-07-25 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Folic acid (Active Comparator): 30 patinets will receive Orally 5mg tablet two times daily for 8 weeks
  Interventions: Drug: Folic Acid Tablet
- Control (Placebo Comparator): 30 patinets will receive Orally 5mg tablet two times daily for 8 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Folic Acid Tablet — oral 5mg tablet two times daily for 8 weeks
  Other Names: Vitamin B-9,Folison
  Arms: Folic acid
Other: Placebo — orally 5mg two times daily for 8weeks
  Arms: Control

SUMMARY:
This is a prospective single center, randomized, double-blind, 2 arm placebo-controlled study in subjects with Parkinson's disease receiving levodopa .The patients will be randomized to receive tablet Folic Acid 10 mg per day or placebo for 8 weeks. The safety and efficacy outcome measures will be assessed at baseline and 8 weeks.

DETAILED DESCRIPTION:
Parkinson's disease is a progressive neurodegenerative disorder that is caused by degeneration of dopaminergic neuron in the substantia nigra. Most commonly used drug, levodopa can improve the dopamine level in brain but levodapa causes hyperhomocysteinmia as a result increse neurotoxicity,oxidative stress and motor fluctuations and dyskinesia in many patients. Folic acid has been reduced homocystein level in levodopa treated Parkinson's disease on animal model and also reduced Levodopa induced dyskinesia without compromising the motor benefits of Levodopa. Therefore, the present study is to attempt to improve the sign symptoms of Parkinson's disease by giving folic acid along with Levodopa.

This study is a Randomized, Double-Blind, Placebo-Controlled Trial and conducting at Department of Pharmacology, BSMMU in collaboration with Department of Neurology, BSMMU. A total of 60 patients suffering from Parkinson's disease is selected according to inclusion and exclusion criteria. The diagnosis of the patients suffering from Parkinson's disease will be performed by a neurologist at movement disorder clinic of department of Neurology, BSMMU. Patients will undergo MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) to assess the severity of the disease. The patients will be randomly allocated into two arms: control and intervention. Patients in intervention arm consisted of 30 patients who will receive levodopa plus folic acid orally for 8 weeks. On the other hand, control arm consisted of 30 patients who will receive levodopa plus placebo for 8 weeks. The severity of Parkinson's disease will be assessed 8 weeks follow up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed PD patients taking levodopa for at least 6months.
* Mild to moderate Parkinson's disease patient according to Hoehn and Yahr staging, stage -I, II, III
* Homocysteine level ≥ 13 µmol/L

Exclusion Criteria:

* Secondary causes of parkinsonism
* Prior stereotactic surgery for PD
* Suffering from active malignancy
* Known hypersensitivity to folic acid
* Multivitamin supplementation within 30 days of enrollment
* Patients taking anticonvulsant, oral contraceptive pill, disease modifying anti-rheumatic drugs
* Pregnancy or lactating mother
* Has any clinically significant medical condition that could interfere with the subject's ability to safely participate in the study or to be followed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-16 (Actual); Primary Completion 2024-07-16 (Estimated); Study Completion 2024-07-16 (Estimated)

PRIMARY OUTCOMES:
Effect of folic acid on motor aspects of daily living in levdopa treated of Parkinson's disease patients | 8 weeks
  Assessing and comparing the severity of symptoms of Parkinson's disease of two groups by using MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) at baseline and 8 weeks following folic acid and placebo supplementation.

SECONDARY OUTCOMES:
Serum homocysteine | 8weeks
  will be measured before and after intervention
Serum malondialdehyde level | 8weeks
  will be measured before and after intervention
Serum glutathion | 8weeks
  will be measured before and after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- BSMMU, Dhaka, Bangladesh